CLINICAL TRIAL: NCT00439114
Title: Comparison of Ultrasonic Pachymetry With Orbscan in Corneal Haze
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Other Study IDs: KA05/207
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2007-02-23 (Estimated); Status verified 2007-02

CONDITIONS: Corneal Opacity
Keywords: Corneal topography, corneal opacity, keratitis, trachoma
MeSH Terms: conditions — Corneal Opacity; Keratitis; Trachoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study is planned to compare the results of ultrasonic and Orbscan pachymetry in corneal haze not related to surgery. Corneal haze is graded with slit-lamp by a single examiner. Ultrasonic and Orbscan II pachymetry measurements are obtained. Paired t and Kruskal-Wallis tests are used to evaluate the difference between ultrasonic and Orbscan pachymetry measurements. Correlation of the two methods and haze grade is determined with Kendall's tau-b correlation analysis.

DETAILED DESCRIPTION:
We planned this study to compare the results of ultrasonic and Orbscan pachymetry in corneal haze not related to surgery. In this institutional based, prospective, controlled clinical trial subjects with corneal haze not related to surgery are included. Normal eyes are used as control group to calculate the customized acoustic factor. Corneal haze is graded with slit-lamp by a single examiner. Ultrasonic and Orbscan II pachymetry measurements are obtained by one technician each masked to the other measurement. Paired t and Kruskal-Wallis tests are used to evaluate the difference between ultrasonic and Orbscan pachymetry measurements. Correlation of the two methods and haze grade is determined with Kendall's tau-b correlation analysis. According to the results of the study, we will determine which method is accurate in subjects with corneal haze.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant corneal haze on slit-lamp are included in the study group. 50 eyes of 50 age-matched patients with normal eye and clear cornea are included in the control group. Only one eye of each subject is included.

Exclusion Criteria:

* Exclusion criteria to participate in the study are previous ocular surgery, history of contact lens use, glaucoma, and topical ocular medication use, excluding artificial tears.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Rana Altan-Yaycioglu, M.D., Principal Investigator — Baskent University, Faculty of Medicine, Department of Ophthalmology
Locations (1):
- Baskent University, Faculty of Medicine, Adana Hospital, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Boscia F, La Tegola MG, Alessio G, Sborgia C. Accuracy of Orbscan optical pachymetry in corneas with haze. J Cataract Refract Surg. 2002 Feb;28(2):253-8. doi: 10.1016/s0886-3350(01)01162-2. PMID 11821206
- [Background] Iskander NG, Anderson Penno E, Peters NT, Gimbel HV, Ferensowicz M. Accuracy of Orbscan pachymetry measurements and DHG ultrasound pachymetry in primary laser in situ keratomileusis and LASIK enhancement procedures. J Cataract Refract Surg. 2001 May;27(5):681-5. doi: 10.1016/s0886-3350(01)00820-3. PMID 11377895
- [Derived] Altan-Yaycioglu R, Pelit A, Akova YA. Comparison of ultrasonic pachymetry with Orbscan in corneal haze. Graefes Arch Clin Exp Ophthalmol. 2007 Dec;245(12):1759-63. doi: 10.1007/s00417-007-0578-5. Epub 2007 Jun 22. PMID 17583820